CLINICAL TRIAL: NCT04407130
Title: Ivermectin and Doxycycline in Combination or Ivermectin Alone for the Treatment of Adult Bangladeshi Patients Hospitalized for COVID-19: a Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: Efficacy and Safety of Ivermectin and Doxycycline in Combination or IVE Alone in Patients With COVID-19 Infection.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR-20039
Record Dates: First submitted 2020-05-17; First posted 2020-05-29 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2020-06

CONDITIONS: COVID-19 Patients
MeSH Terms: interventions — Ivermectin; Doxycycline

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tab Ivermectin +Cap Doxycycline (Active Comparator): 200 mcg/kg (12 mg tablet) ivermectin (IVERA) single dose and 200 mg stat doxycycline day-1 followed by 100mg doxycycline 12hrly for 4 day (i.e. day2-day5)
  + Placebo one tablet D2-5
  Interventions: Drug: Ivermectin + Doxycycline + Placebo
- Tab Ivermectin (Active Comparator): Ivermectin - 200 mcg/kg (12 mg tablet) once per day D1-D5
  + Placebo two tablets D1 followed by Placebo one tablet D2-5
  Interventions: Drug: Ivermectin + Placebo
- Placebo (Placebo Comparator): Drug: Placebo
  3 Placebo tablets D1 followed by 2 tablets D2-5
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ivermectin + Doxycycline + Placebo — Arm I: 200 mcg/kg (12 mg tablet) ivermectin (IVERA) single dose and 200 mg stat doxycycline day-1 followed by 100mg doxycycline 12hrly for 4 day (i.e. day2-day5)
  Placebo one tablet D2-5
  Other Names: Tab IVERA +Cap Doxycycline
  Arms: Tab Ivermectin +Cap Doxycycline
Drug: Ivermectin + Placebo — Arm II: Ivermectin - 200 mcg/kg (12 mg tablet) once per day D1-D5 + Placebo two tablets D1 followed by Placebo one tablet D2-5
  Other Names: Tab IVERA
  Arms: Tab Ivermectin
Drug: Placebo — Arm III: 3 Placebo tablets D1 followed by 2 tablets D2-5
  Other Names: Tab Placebo
  Arms: Placebo

SUMMARY:
Burden:

Initial outbreak of corona virus disease 2019 (COVID-19) was reported from Wuhan, China in early December 2019.Presently known to be caused by a novel beta-corona virus, named as Severe acute respiratory syndrome corona virus 2 ( SARS-CoV-2).

World Health Organization (WHO) declared a pandemic on March.

The clinical characteristics of COVID-19 include respiratory symptoms, fever, cough, dyspnoea and pneumonia

Infected individuals exhibit:

1. Mostly mild illness (80% +) recover without any treatment (~80%)
2. Moderate illness that needs hospitalization and recovers after standard
3. supportive treatment (~14%)
4. Critical illness (~5%) needs ICU support
5. Death (1-2% )

COVID-19 has now spread >210 countries and territories globally. SARS-CoV-2 is a respiratory virus which spreads primarily through droplets generalized when an infected person coughs or sneezes or through droplets of saliva or discharge from the nose.

Symptomatic management remains the mainstay of treatment strategy. Mortality appears to be more common in older individuals and those with co-morbidities, such as chronic lung disease, cardiovascular disease and diabetes. Young people with no comorbidities also appear to be at risk for critical illness including multi-organ failure and death. Seen more in Bangladesh between 21-40 yrs of age.

Knowledge Gap:

There is no specific treatment against this new virus that WHO has officially declared until now.There are many pharmacologic therapies that are being used or considered for treatment of COVID-19. National Guidelines on Clinical Management of Corona virus Disease 2019 (Covid-19): V 5.0 date 9th April 2020) CDC, DGHS, GoB

Thus an RCT is urgently needed in Bangladesh: Based on recent literatures on Rx studies in COVID-19 patients from other countries as well as its availability & affordability of those repurposed medicines

DETAILED DESCRIPTION:
Objectives:

General Objective:

The aim of the study is to evaluate efficacy and safety of ivermectin in combination with doxycycline or ivermectin alone for the treatment of hospitalized SARS-CoV-2 infected adult Bangladeshi COVID-19 +ve patients and to compare with placebo; where all three arms will receive the standard care of treatment of COVID-19 infected patients in the hospital. By successful demonstration of the safety and efficacy of these repurposed medicines, it may have the potential to play an important role in the treatment of COVID-19+ve patients.

Specific Objective:

1. Duration of the virological clearance rate
2. Days required for remission of fever and cough

Secondary Objective:

* Patients requiring oxygen
* Patients failing to maintain SpO2 >88 despite oxygenation
* Number of days on oxygen support
* Chest X-ray improvement
* Duration of hospitalization
* All cause mortality

ELIGIBILITY:
Inclusion criterion:

* Bangladeshi aged 18-65 years admitted to any of the aforementioned study sites (hospitals)
* Either sex
* At the enrollment having at least one of the following symptoms: Temp 37.5 C or above, Cough, Sore throat
* SpO2 >94%
* Duration of illness ≤ 7 days
* No oxygen support on enrollment
* Capable of swallowing oral medication
* PCR positive for SARS-CoV2 virus
* The participant properly informed about the study and agreed to sign the informed consent form (ICF)

Exclusion Criteria:

* Allergy to ivermectin or doxycycline; or other contraindications to any of the study medications
* History of chronic heart disease (IHD, heart failure, documented cardiomyopathy etc)
* History of chronic liver disease (SGPT value more than 3 times of normal value)
* History of chronic kidney disease (S. Creatinine for male >1.3 mg/dL or >115 µmol/L and for female >1.2 mg/dL or >106.1 µmol/L)
* Pregnant or lactating women
* Participated in any other clinical trial within last 4 weeks
* H/o received Ivermectin/Doxycycline within last 7 days

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Virological clearance | within 7 days after enrollment
  • Presence of virus will be negative on Day 7 detected by RT PCR
Remission of fever | within 7 days after enrollment
  • Body temperature will be < 37.5 C by day 7 detected by Infrared thermometer
Remission of cough | within 7 days after enrollment
  • Remission of cough: No signs of cough showing respiratory rate within 12-20/ min, on day7

SECONDARY OUTCOMES:
Patients requiring oxygen | within 7 days after enrollment
  Detected SPO2 level <94% on Day 7or before by pulse oxymeter
Patients failing to maintain SpO2 >93% despite oxygenation | within 7 days after enrollment
  Patients who fail to maintain pulse oxymeter detected SpO2 level>93% despite O2 supplementation of 2-6 L/min, on Day 7 or before
Number of days on oxygen support | within 7 days after enrollment
  Any number of days on oxygen support on Day 7 or before recorded in CRF
Duration of hospitalization | within 14 days after enrollment
  Hospital stay ≥7days to ≤14 days as per CRF records
All causes of mortality | within 14 days after enrollment
  Death any time during 14 days of study period from any cause recorded in CRF and Hospital death certificate

CONTACTS AND LOCATIONS:
Overall Officials: Wasif Ali Khan, MBBS, MHS, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Icddr,B, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No